CLINICAL TRIAL: NCT04592692
Title: A Pharmacokinetic and Clotting Activity Study of FVIII-PEGLip Administered Intravenously to Severe Haemophilia A Patients With and Without Inhibitors to FVIII
Brief Title: A Pharmacokinetic and Clotting Activity Study of FVIII-PEGLip
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ascension Healthcare Development Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-SelectAte-II-01
Record Dates: First submitted 2020-09-21; First posted 2020-10-19 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Hemophilia A With Inhibitor
Keywords: Hemophilia A; Inhibitors
MeSH Terms: conditions — Hemophilia A | interventions — simoctocog alfa (Nuwiq)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Inhibitors (Experimental): Patients with inhibitors to FVIII
  Interventions: Drug: PEGylated Liposome (PEGLip)
- Non-inhibitors (Other): Patients without inhibitors to FVIII
  Interventions: Drug: PEGylated Liposome (PEGLip)

INTERVENTIONS:
Drug: PEGylated Liposome (PEGLip) — Intravenous co-administration of PEGLip with Simoctocog alfa
  Other Names: Simoctocog alfa

SUMMARY:
The purpose of this study is to demonstrate that PEGylated liposomes (PEGLip) can shield FVIII from the immune system and inhibitors, and therefore provide a prophylactic FVIII replacement therapy for patients with inhibitors to FVIII.

DETAILED DESCRIPTION:
This is an open-label multicenter trial for patients with severe haemophilia A with inhibitors to FVIII and without inhibitors as control. The trial consists of 4 periods: Screening, Stage A, Stage B and Safety Follow-up.

After signing informed consent, patients are assessed for eligibility during a Screening period lasting up to 21 days.

All eligible patients enter Stage A - Regimen estimation. The non-inhibitor patients receive a single IV injection at a dose of 35 IU/kg FVIII reconstituted with Water For Injection. Following a 4-day wash-out period, these patients as well as patients with inhibitors receive a single IV injection of FVIII-PEGLip at a dose of 35 IU/kg FVIII + PEGLip 22 mg/kg to determine the duration of haemostatic cover and therefore required injection frequency to prevent bleeds.

Stage B - multiple dosing: all patients receive injections of FVIII-PEGLip for 6 weeks at a frequency determined in Stage A for each individual patient.

Safety follow-up: 15 and 30 days after the last injection of FVIII-PEGLip, patients are contacted for any adverse events or bleeding episodes.

ELIGIBILITY:
Inclusion Criteria:

* Male adult patients aged 18 to 60 years;
* Severe Haemophilia A (FVIII plasma level <1IU/dL) with documented history of bleeds (for at least 6 months prior to enrolment);
* For patients without inhibitors: inhibitor titre < 0,6 Bethesda units and no medi-cal history of inhibitors;
* For patients with inhibitors: inhibitor titre ≥0,6 Bethesda units or documented medical history of inhibitors titre ≥0,6 Bethesda units;
* Adequate hematologic function, defined as platelet count ≥ 100,000/μL and hemoglobin ≥ 8 g/dL (≥ 4.97 mmol/L) at the time of screening;
* Adequate hepatic function, defined as total bilirubin ≤ 1.5 × the upper limit of normal (ULN) (excluding Gilbert's syndrome) and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 ×ULN at the time of screening; no clinical signs or known laboratory/radiographic evidence consistent with cirrho-sis;
* Adequate renal function, defined as serum creatinine ≤ 2.5 × ULN and creati-nine clearance by Cockcroft-Gault formula ≥ 30 mL/min;
* Patient's written informed consent, confirming his willingness to comply with the requirements of this protocol.

Exclusion Criteria:

* Low platelet counts (<100000 / μl);
* Congenital or acquired bleeding defects (including acquired hemophilia) other than Hemophilia A;
* Abnormal renal function (serum creatinine concentrations greater than 1.3 mg/dL);
* Active hepatic disease (persistent aspartate aminotransferase [AST] or alanine aminotransferase [ALT] increases to greater than five times the upper limit of normal);
* A history of severe adverse reactions to blood products and/or plasma derived FVIII concentrates or liposomes, or PEG, or Nuwiq;
* A history of allergic reactions to bypassing agents;
* Any concomitant immunological disease (e.g. autoimmune chronic active hepati-tis, autoimmune thrombocytopenic purpura or Immune Thrombocytopenic Pur-pura (ITP), lupus, Multiple Sclerosis (MS));
* Patients receiving immunosuppressive treatment (excluding glucocorticoids);
* Patients receiving therapy with interferon;
* Patients receiving any immune tolerance induction (ITI) therapy at the moment of the screening;
* Any individual with known dyslipidemia disease or actively taking cholesterol lowering drugs for the treatment of hypercholesterolemia or hyperlipidemia (e.g., statins, cholesterol absorption inhibitors, bile acid sequestrates, nicotinic acid or fibrates);
* Intake of NSAIDs (except COX-2 inhibitors), acetylsalicylic acid (Aspirin) or any other antiplatelet agents, opioids.;
* Patients who have participated in another Clinical Trial (including medical device studies) within the past 60 days;
* Concurrent disease, treatment, or abnormality in clinical laboratory tests that could interfere with the conduct of the study or that would, in the opinion of the investigator or Sponsor, preclude the patient's safe participation in and completion of the study or interpretation of the study results, according to the Investigator.
* For patients without inhibitors - a history of demonstrating long half-lives for FVIII.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male patients only
Enrollment: 20 (Estimated)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Clotting activity based on ROTEM [single dose] | 7 days
  Clotting profile of single IV injection of FVIII-PEGLip based on key ROTEM parameters (CT+CFT) determined at 0 hours (pre-injection) and at 20 min, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144 and 168 hours after injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Clotting activity based on FVIII:C concentration [single dose] | 7 days
  Clotting profile of single IV injection of FVIII-PEGLip based on FVIII:C plasma assay measured at 0 hours (pre-injection) and at 20 min, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144 and 168 hours after injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Clotting activity based on ROTEM [multiple dose] | 6 weeks
  Dynamics of blood clotting activity as quantified by key ROTEM parameters (CT+CFT) measured before and 20 minutes after each injection of FVIII-PEGLip at weeks 2, 4 and 6 of 6-week multiple dosing of FVIII-PEGLip in severe Haemophilia A patients with inhibitors and patients without inhibitors.
Bleed frequency | 6 weeks
  Frequency of spontaneous bleeding episodes and average length (days) of bleeding-free periods
Area under the concentration-time curve (AUC) of FVIII:C (FVIII-PEGLip) [single dose] | 7 days
  AUC0-∞ of FVIII:C after single IV FVIII-PEGLip injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Area under the concentration-time curve (AUC) of FVIII:C (FVIII-WFI) [single dose] | 4 days
  AUC0-∞ of FVIII:C after single IV FVIII-WFI injection in severe Haemophilia A patients without inhibitors
Maximum plasma concentration (Cmax) of FVIII:C (FVIII-PEGLip) [single dose] | 7 days
  Cmax of FVIII:C after single IV FVIII-PEGLip injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Maximum plasma concentration (Cmax) of FVIII:C (FVIII-WFI) [single dose] | 4 days
  Cmax of FVIII:C after single IV FVIII-WFI injection in severe Haemophilia A patients without inhibitors
Time to reaching maximum plasma concentration (Tmax) of FVIII:C (FVIII-PEGLip) [single dose] | 7 days
  Tmax of FVIII:C after single IV FVIII-PEGLip injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Time to reaching maximum plasma concentration (Tmax) of FVIII:C (FVIII-WFI) [single dose] | 4 days
  Tmax of FVIII:C after single IV FVIII-WFI injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Half-life (t1/2) of FVIII:C (FVIII-PEGLip) [single dose] | 7 days
  T1/2 of FVIII:C after single IV FVIII-PEGLip injection in severe Haemophilia A patients with inhibitors and in patients without inhibitors
Half-life (t1/2) of FVIII:C (FVIII-WFI) | 4 days
  T1/2 of FVIII:C after single IV FVIII-WFI injection in severe Haemophilia A patients without inhibitors

SECONDARY OUTCOMES:
Inhibitor titres | Approximately 12 weeks
  Individual changes of inhibitor titres from baseline measurement to 168 hours after single IV injection of FVIII-PEGLip and at weeks 2, 4, and 6 of 6-week FVIII-PEGLip multiple dosing period
Area under the concentration-time curve (AUC) of PEGLip [single dose] | 7 days
  AUC0-∞ of PEGLip determined at 0 hours (pre-injection) and at 20 min, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144 and 168 hours after single IV injection of FVIII-PEGLip
Maximum plasma concentration (Cmax) of PEGLip [single dose] | 7 days
  Cmax of PEGLip determined at 0 hours (pre-injection) and at 20 min, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144 and 168 hours after single IV injection of FVIII-PEGLip
Time to reaching maximum plasma concentration (Tmax) of PEGLip [single dose] | 7 days
  Tmax of PEGLip determined at 0 hours (pre-injection) and at 20 min, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144 and 168 hours after single IV injection of FVIII-PEGLip
Half-life (t1/2) of PEGLip [single dose] | 7 days
  t1/2 of PEGLip determined at 0 hours (pre-injection) and at 20 min, 1, 2, 4, 8, 24, 48, 72, 96, 120, 144 and 168 hours after single IV injection of FVIII-PEGLip
PEGLip concentration [multiple dose] | 6 weeks
  PEGLip concentration measured before and 20 minutes after each injection of FVIII-PEGLip at weeks 2, 4 and 6 of 6-week multiple dosing of FVIII-PEGLip

OTHER OUTCOMES:
Adverse events | Approximately 12 weeks
  Adverse events / Serious Adverse Events developed in the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sam Yurdakul, Study Director — Ascension Healthcare
Locations (5):
- Russia (5):
  - Kemerovo District Clinical Hospital, Kemerovo
  - Kirov Scientific Research Institute of Hematology and Blood Transfusion, Kirov
  - National Medical Research Centre of Hematology, Moscow
  - Novosibirsk State Medical University, Novosibirsk City Haematology Center, Novosibirsk
  - Samara State Medical University, Samara

IPD SHARING:
Plan to Share IPD: No